CLINICAL TRIAL: NCT06103123
Title: MYocarditis and/or Pericarditis Following mRNA COVID-19 VACCination National Surveillance Study
Acronym: MYCOVACC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cardiology Research UBC (Other)
Responsible Party: Sponsor
Other Study IDs: MYCOVACC
Record Dates: First submitted 2023-05-29; First posted 2023-10-26 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Myocarditis; Myocarditis Acute; Pericarditis; Pericarditis Acute
MeSH Terms: conditions — Myocarditis; Pericarditis | interventions — Magnetic Resonance Imaging; Caves

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- mRNA COVID-19 vaccine associated myocarditis: Participants who had developed myocarditis within 42 days of getting a mRNA COVID-19 vaccine
  Interventions: Diagnostic Test: Stand of care ECG, Holter, MRI, ECHO, Quality of life questionnaire
- mRNA COVID-19 vaccine associated pericarditis: Participants who had developed pericarditis within 42 days of getting a mRNA COVID-19 vaccine
  Interventions: Diagnostic Test: Stand of care ECG, Holter, MRI, ECHO, Quality of life questionnaire
- COVID-19 infection associated myocarditis: Participants who had developed myocarditis within 42 days of being infected with the SARS-COV-2 virus
  Interventions: Diagnostic Test: Stand of care ECG, Holter, MRI, ECHO, Quality of life questionnaire
- COVID-19 infection associated pericarditis: Participants who had developed pericarditis within 42 days of being infected with the SARS-COV-2 virus
  Interventions: Diagnostic Test: Stand of care ECG, Holter, MRI, ECHO, Quality of life questionnaire
- Alternative etiology myocarditis: Any participants with myocarditis that is not associated with the mRNA COVID-19 vaccine or SARS-COV-2 viral infection
  Interventions: Other: Baseline Quality of Life questionnaire

INTERVENTIONS:
Diagnostic Test: Stand of care ECG, Holter, MRI, ECHO, Quality of life questionnaire — Stand of care ECG, Holter, MRI, ECHO, Quality of life questionnaire will be used to follow the clinical outcomes and patient reported outcomes to assess for study objectives
  Groups: COVID-19 infection associated myocarditis; COVID-19 infection associated pericarditis; mRNA COVID-19 vaccine associated myocarditis; mRNA COVID-19 vaccine associated pericarditis
Other: Baseline Quality of Life questionnaire — Only baseline quality of life questionnaires will be utilized in the alternative etiology myocarditis cohort as they will not be followed up in the study
  Groups: Alternative etiology myocarditis

SUMMARY:
Myocarditis is inflammation of the heart muscle. Pericarditis is inflammation of the lining surrounding the heart muscle. Symptoms of these conditions can include pain in the chest and rapid or irregular heartbeat. There are many different causes for myocarditis and pericarditis including COVID-19 infection.

The MYCOVACC study will identify patients using local screening strategies, including research communications, care provider referrals, and medical record review. The retrospective component of the study will collect information about patients suffering from vaccine associated myopericarditis and COVID-19 associated myopericarditis. Consenting patients will then be prospectively followed according to standard of care protocols. The main objectives of MYCOVACC are to describe the rate of major adverse cardiovascular events, functional outcomes including quality of life, and myocardial recovery through imaging.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for vaccine associated myocarditis/pericarditis.

  1. COVID-19 vaccination within previous 42 days. AND
  2. At least one cardiac symptom of suspected myocarditis/pericarditis (Appendix 5).

     OR At least two non-specific symptoms (Appendix 5). OR In infants and young children, at least two non-specific pediatric symptoms (Appendix 5).

     OR No symptoms, but abnormal histopathology or a combination of abnormal cardiac biomarkers with abnormal cardiac imaging (echo or MRI).

     AND
  3. At least one of the following objective findings (Brighton Criteria case definitions, Appendices 1 to 5):

     1. Histopathologic examination of myocardial tissue (autopsy or endomyocardial biopsy) showed myocardial inflammation.
     2. Elevated myocardial biomarker (Troponin T, Troponin I, or CK-MB).
     3. Cardiac MRI abnormality.
     4. Echocardiographic abnormality.
     5. New or worsening arrhythmia on electrocardiogram, Holter monitor, or telemetry.
     6. Elevated inflammation biomarkers: erythrocyte sedimentation rate (ESR), C-reactive protein (CRP), hs-CRP, or D-Dimer.
     7. Physical examination pericardial friction rub or pulsus paradoxus.
     8. Pericardial fluid or inflammation by imaging (echo, MRI, or CT).
     9. Enlarged heart on chest radiograph.

     AND
  4. No alternative cause of presentation. e.g. infectious or autoimmune myocarditis.
* Inclusion criteria for COVID-19 associated myocarditis/pericarditis

  1. COVID-19 infection within the previous 42 days.

     AND
  2. Myocarditis/pericarditis as per Brighton Criteria for vaccine associated myocarditis/pericarditis.

     AND
  3. No alternative cause of presentation.

Inclusion criteria alternative etiology myocarditis.

1. Myocarditis/pericarditis as per Brighton Criteria for vaccine associated myocarditis/pericarditis.

   AND
2. No alternative cause of presentation.

Exclusion Criteria:

* For prospective invitation and follow-up, inability to provide informed consent. Consent will be sought from patients or their authorised substitute decision maker.
* Patients not fulfilling Brighton Criteria levels 1-3 will be excluded if they are level 4 (insufficient evidence for myocarditis) or Level 5 (not myocarditis) or have an alternative diagnosis such as myocardial infarction.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who have suffered or are suffering from 1) COVID-19 infection associated myocarditis, 2) COVID-19 infection associated pericarditis, 3) COVID-19 vaccine associated myocarditis, 4) COVID-19 vaccine associated pericarditis, 5) Alternative etiology myocarditis, 6) Alternative etiology pericarditis
  Definition of myocarditis and pericarditis follows standard clinical definition as outlined in "Brighton Collaboration myocarditis case definition and levels of diagnostic certainty 1,2 and 3"
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-04-23 (Actual); Primary Completion 2025-03-23 (Estimated); Study Completion 2025-04-23 (Estimated)

PRIMARY OUTCOMES:
Composite Major Adverse Cardiac Event (MACE) at 30 days post vaccination (preferred by cardiovascular community) and at 42 days post vaccination (preferred by vaccine monitoring investigators) | From date of vaccination and up to 3 years
  Including any of:
  * Death from any cause.
  * Ventricular arrhythmia (ventricular fibrillation or ventricular tachycardia).
  * Heart block (type II or type III block).
  * Heart failure (national guideline criteria).
  * Left ventricular systolic dysfunction (left ventricular ejection fraction [LVEF] <55%).
  * Cardiac tamponade.
Recovery of cardiac function in patients with previously documented abnormal cardiac function | Through study completion, an average of 3 years
  Patients with Left Ventricular Ejection Fraction (LVEF)<55% during anytime at baseline, with LVEF increase by 5% from worst baseline measurement
Quality of life using validated instruments at baseline, 3 months, 12 months, and annually | Through study completion, an average of 3 years
  Quality of life: EQ-5D-5L questionnaire for adults or EQ-5D-Y questionnaire for children.
Depression and anxiety using validated instruments at baseline, 3 months, 12 months, and annually | Through study completion, an average of 3 years
  Depression and anxiety data: PHQ-9 and GAD-7.
Physical activity using validated instruments at baseline, 3 months, 12 months, and annually | Through study completion, an average of 3 years
  Physical activity: International Activity Questionnaire.

SECONDARY OUTCOMES:
Individual components of primary composite endpoint at 30 days and 42 days post mRNA COVID-19 vaccination? | From date of vaccination for up to three years
Rate of atrial arrhythmias after mRNA COVID-19 vaccination? | From date of vaccination for up to three years
Rate of all-cause and cardiovascular mortality after mRNA COVID-19 vaccination? | From date of vaccination for up to three years
Rate of all-cause and cardiovascular hospitalization after mRNA COVID-19 vaccination? | From date of vaccination for up to three years
Rate of recurrence of myocarditis/pericarditis after mRNA COVID-19 vaccination? | From date of vaccination for up to three years
Rate of constrictive pericarditis after mRNA COVID-19 vaccination? | From date of vaccination for up to three years

CONTACTS AND LOCATIONS:
Overall Officials: Nathaniel Hawkins, MD, Principal Investigator — Vancouver General Hospital
Locations (1):
- Vancouver General Hospital, Vancouver, British Columbia, Canada

REFERENCES:
- See also: Related Info — https://ccs.ca/mycovacc/

DOCUMENTS (1):
  • Study Protocol (2023-04-12): https://cdn.clinicaltrials.gov/large-docs/23/NCT06103123/Prot_000.pdf